CLINICAL TRIAL: NCT04001036
Title: Efficacy and Safety Assessments of a Peritoneal Dialysis Solution Containing Glucose, Xylitol and L-Carnitine Compared to Standard PD Solutions in Continuous Ambulatory Peritoneal Dialysis (CAPD)
Brief Title: Efficacy and Safety Assessments of a Peritoneal Dialysis Solution Containing Glucose, Xylitol, and L-Carnitine in CAPD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: prematurely interrupted due to significant difficulties in the completion of the sample size defined by the study protocol
Sponsor: Iperboreal Pharma Srl (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP-001-09
Record Dates: First submitted 2019-06-26; First posted 2019-06-27 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2022-08

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Xylitol; Glucose; Carnitine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental peritoneal dialysis solution IPX15 (Experimental): Patients will receive treatment with the experimental solution for nocturnal (long-dwell) exchange. For daily (short-dwell) exchanges, all patients will continue the 1 to 3 bags of glucose peritoneal dialysis solution as for their pre-randomization prescription.
  Interventions: Drug: 1.5% Xylitol, 0.5% Glucose, and 0.02% L-carnitine
- Experimental peritoneal dialysis solution IPX07 (Experimental): Patients will receive 1 to 3 daily (short-dwell) exchanges with the experimental solution (the number of exchanges will be based on their pre-randomization prescription). All patients will receive icodextrin for nocturnal (long-dwell) exchange.
  Interventions: Drug: 0.7% Xylitol, 0.5% Glucose, and 0.02% L-carnitine

INTERVENTIONS:
Drug: 1.5% Xylitol, 0.5% Glucose, and 0.02% L-carnitine — One bag for nocturnal (long-dwell) exchange.
  Other Names: IPX15
  Arms: Experimental peritoneal dialysis solution IPX15
Drug: 0.7% Xylitol, 0.5% Glucose, and 0.02% L-carnitine — One to three, daily (short-dwell) exchanges
  Other Names: IPX07
  Arms: Experimental peritoneal dialysis solution IPX07

SUMMARY:
Prospective, randomized, controlled clinical trial. The aim is to compare the effects of the peritoneal dialysis solution IPX15, containing glucose (0.5%), xylitol (1.5%) and L-carnitine (0.02%) as osmotic agents (comparable to the standard 2.5% glucose PD solution), for the nocturnal exchange with the PD solution IPX07, containing glucose (0.5%), xylitol (0.7%) and L-carnitine (0.02%) as osmotic agents (comparable to the standard 1.5% glucose PD solution), for the diurnal (short dwell) exchanges. Planned total recruitment is 40 patients with stable end-stage renal disease (ESRD) treated by continuous ambulatory peritoneal dialysis (CAPD). Treatment duration will be 4 weeks plus a 4 weeks safety follow up with no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ESRD treated for at least three months with CAPD, as stated by the medical staff of the center;
* Stable clinical condition within four weeks before the screening period, certified by medical/surgical history, physical examination and laboratory exploration;
* Hemoglobin level ≥ 9g/dL;
* Absence of acute peritonitis and/or peritoneal catheter infection (either exit site or subcutaneous tunnel) episodes within three months before selection;
* To understand and sign an informed consent form.

Exclusion Criteria:

* History of alcohol or drug abuse in the last six months before selection for the study;
* Androgen therapy in the last six months before selection;
* Active infections;
* History of congestive heart failure stage III and IV New York Heart Association (NYHA);
* History of major cardiovascular events like stroke, acute myocardial infarction, coronary or other arterial revascularization procedures in the last three months before selection;
* Clinically relevant cardiac arrhythmia;
* Clinically relevant abnormalities of functional hepatic tests;
* Therapy with L-carnitine or its derivatives in the last three months before selection;
* Pregnancy, lactating women or female subjects of childbearing potential who do not use an effective method of contraception;
* Presence of relevant chronic medical conditions that could suggest exclusion of patient from the study or could interfere with the assessment of study parameters, especially if the life expectancy is less then one year;
* Participation in another clinical study within the past month;
* Known allergic reactions to L-carnitine or xylitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Daily ultrafiltration volume | 28 days
  Change from baseline

SECONDARY OUTCOMES:
Peritoneal equilibration test | 28 days
  Change from baseline
Weekly total urea Kt/V | 28 days
  Change from baseline
Weekly total creatinine clearance | 28 days
  Change from baseline
Adverse Events | 2 months
  Information about all adverse events, whether volunteered by the patient, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, will be collected, recorded and followed as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Bonomini, MD, Principal Investigator — Institute of Nephrology, G. D'annunzio University, Chieti, Italy
Locations (1):
- Department of Nephrology, University of Chieti, Chieti, Italy

REFERENCES:
- [Derived] Nishioka N, Luo Y, Taniguchi T, Ohnishi T, Kimachi M, Ng RC, Watanabe N. Carnitine supplements for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013601. doi: 10.1002/14651858.CD013601.pub2. PMID 36472884